CLINICAL TRIAL: NCT07227935
Title: Sustaining Quality Physical Education for Healthy Kids
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Weiyun Chen, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00241100
Record Dates: First submitted 2025-10-19; First posted 2025-11-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Smart-Quality Physical Education
Keywords: Quality Physical Education, Heart Zone Moves System

STUDY DESIGN:
Intervention Model Description: During the Smart-Quality Physical Education (PE) intervention, the PE teacher will integrate the Heart Zone Moves System into teaching each PE lessons, where students will wear the heart rate monitor on his/her forearm to self-monitor his/her real time engagement in moderate-to-vigorous physical activity (MVPA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smart-Quality Physical Education (Experimental): For the Smart-Quality Physical Education (Smart-QPE) intervention, PE teachers integrates the Heart Zone Moves System into teaching quality physical education lessons. During the Smart-QPE lessons, students wear the heart rate monitors synced to system to self-monitor their heart rates corresponding to light, moderate, and vigorous intensity physical activity.
  Interventions: Behavioral: Smart-QPE

INTERVENTIONS:
Behavioral: Smart-QPE — During the Smart-QPE intervention spanning in October - November, 2025, the physical education teacher integrate the Heart Zone Moves System into teaching quality physical education lessons; students wear the heart rate monitor on his/her forearm to self-monitor his/her real time engagement in moderate-to-vigorous physical activity (MVPA) to maximize students MVPA time.

SUMMARY:
The purpose of the study is to examine the effects of the technology-enhanced quality physical education (Smart-QPE) lessons on physical activity, cardiorespiratory fitness, social emotional learning (SEL) skills, and mental well-being in school students.

DETAILED DESCRIPTION:
Students in 4th-7th grades from 17 elementary and middle schools in Michigan are invited to participate in the study. Students will be assessed with cardiorespiratory fitness, social emotional learning skills, physical activity, and mental well-being at a baseline and the post-intervention tests before and after the Smart-QPE intervention. The Smart-QPE intervention include that PE teachers integrate the Heart Zone Moves System into their teaching quality physical education lesson in October and November, 2025.

ELIGIBILITY:
Inclusion Criteria:

* students are 4rd-7th grade students aged 8-14 years old;
* enroll in the school offered physical education classes;
* being able to read and write in English;
* students can skip any questions they don't want to answer as they respond to the survey questions at the baseline and the post-intervention; and
* students can stop the aerobic fitness test at the baseline and the post-intervention

Exclusion Criteria:

1. students cannot complete the survey, which means that students had difficulty understanding the meaning of each item due to severe cognitive impairment informed by the school nurse/social worker,
2. students do not submit the survey on time (within a week),
3. if a student only submit one survey either at baseline or at the post-intervention,
4. students cannot take the aerobic fitness test, which means that students had difficulty moving their body due to severe physical impairment informed by school nurse/social worker.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — All students including boys and girls and self-identified genders were invited to participate.
Enrollment: 970 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity (MVPA) | During the Smart-QPE intervention period (up to two months).
  The MVPA during the Smart-QPE lessons will be objectively measured by using the Heart Zone Moves System, which is synced to each student's heart rate monitor wore on their forearms.
PACER test | Baseline test and post-intervention test (up to 4 months).
  The PE teacher will administer the PACER test to students for measuring their cardiorespiratory fitness will be assessed during a regular PE lesson.

SECONDARY OUTCOMES:
Assessing Social Emotional Learning Skills Questionnaire | Baseline and post-intervention test (up to 4 months).
  Students' social emotional learning skills will be assessed by completing the Qualtrics Survey. This is online platform survey includes this social emotional learning outcome.
The Physical Activity Questionnaire for Children | Baseline and post-intervention test (up to 4 months).
  Students will complete the Qualtrics Survey, including Physical Activity Questionnaire for Children. Students will respond to 7 items describing a specific setting to engage in physical activity on 5 point-rating scale.
Mental Health and Well-Being questionnaire | Baseline and post-intervention test (up to 4 months).
  Students will complete the Qualtrics Survey, including mental health and mental well-being questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Kinesiology, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
In the IRB-approved consent form, we did not indicate that we will share IPD with other researchers.